CLINICAL TRIAL: NCT02865083
Title: The Effect of a Self-Retaining Pannus Retractor in Obese Patients Undergoing Cesarean Section
Acronym: Traxi
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to reach enrollment goal
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jennifer Goldkamp, MD, MD, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 26533
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Obese Patients Undergoing Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): Subjects will receive use of the Traxi pannus retractor when undergoing cesarean section
  Interventions: Device: Traxi Pannus Retractor
- Standard (No Intervention): Patients will receive use of the standard of care option which is the montgomery straps

INTERVENTIONS:
Device: Traxi Pannus Retractor — traxi® Panniculus Retractor is a retraction device used for retraction of the panniculus during surgical procedures. traxi retracts and holds the panniculus for the duration of the operation, freeing the surgeons hands and those of the staff to better care for the patient.
  Arms: Treatment

SUMMARY:
The purpose of this study is to investigate the effects of the Traxi Pannus retractor in obese patients (BMI ≥30 kg/m2) who undergo Cesarean sections compared to routine pannus retraction techniques. Patients will be randomized to the use of the Traxi retractor during Cesarean section (treatment group) or the use of traditional pannus retraction techniques (control group). The primary outcome to be followed is surgical site disruption. The investigators will also assess the duration of surgery or length of time from skin incision to delivery of the infant, change in hemoglobin, estimated blood loss, postoperative length of stay, need for hospital readmission or emergency room visits, or other complication rates between the two groups.

DETAILED DESCRIPTION:
Surgical site infections (SSI) are an important cause of morbidity following cesarean sections. The rate of surgical site infections following cesarean section in the United States is estimated between 3-15%, depending on the population studied, definitions of surgical site infection used, and length of time studied and is often underestimated. Morbidities include longer length of hospital stay, hospital readmission, wound opening and re-exploration, need for home health care, increased health care costs and loss of productivity. The risk of developing a SSI after a Cesarean section is increased with certain patient characteristics, such as obesity and duration of surgery and is decreased with the use prophylactic antibiotics prior to the skin incision.

Obesity is a significant public health problem and the incidence continues to increase in the United States. It has been shown to be associated with increased risk of SSI after cesarean section in several studies. Olsen et al reviewed 1,605 patients who underwent cesarean section and found increased BMI at admission was an independent risk factor for SSI. In another study of 19,416 women in Israel who had cesarean deliveries, women who had a BMI ≥30 kg/m2 had an increased risk for infection (odds ratio [OR} =2.2; 95% Confidence Interval [CI]. Leth, et al. also found obesity as a risk factor associated with wound infection. In this study of 2,492 consecutive women who had cesarean sections in Denmark, infection rates increased with increasing BMI, with women with a BMI kg/m2 30.0-34.9 having an infection rate of 19.1% and women with a BMI of 35.0-39.9 kg/m2 and of ≥40 kg/m2 both having infection rates of 31.1%. Hypotheses for the increased rate of wound infections in obese patients include decreased vascularity of adipose tissue, increase in wound area, and poorer penetration of prophylactic antibiotics to adipose tissue. Adequate surgical exposure and good visualization are paramount in abdominal surgery. Retraction of the pannus cephalad is often required for adequate visualization and access to the lower abdomen and thus the lower uterine segment. Several studies have been shown that pfannensteil or joel-cohen incisions are superior to vertical incisions due to increased risk of classical cesarean delivery in the case of the obese gravida. Limited studies have been completed to assess supra umbilical incisions.

Other methods of pannus retraction are currently utilized in obstetrics surgery, mostly with surgical tape or Montgomery straps. However, there are currently no clinical trials comparing types of pannus retractors. Potential benefits from the Traxi retractor are decreased operating time, decreased need for additional operating room personnel, and increased ease of delivery of neonate. In addition, the Traxi is designed to stay on for 24 hours in order to elevate the pannus, this will decrease exposure to moisture and possibly other bacteria as the skin begins to heal.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a BMI greater than or equal to 30 kg/m squared, aged 14-50 years old, undergoing non-emergent cesarean section for delivery and require pannus displacement for surgery.

Physicians Inclusion would include any physician who routinely perform C-sections

Exclusion Criteria:

* Patients undergoing emergency Cesarean-section Pre-existing concurrent infection including chorioamnionitis State of immunosuppression (ie. HIV, cancer) Long-term steroid use (>2 days) Patients with a BMI <30 kg/m2, or those with a BMI >/=30kg who do not require pannus retraction.

If there is a rash in the area of retraction Adhesive/tape allergy. Physicians exclusion would include any physician who does not routinely perform C-sections.

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goldkamp, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Standard
Started | 3 | 1
Completed | 0 | 0
Not Completed | 3 | 1
Not completed — Early Termination | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Standard | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] — Data were not collected Population: data were not collected
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Wound Disruption Rates
Description: To determine if there is a difference in wound disruption rates, in obese patients who have Cesarean sections when the Traxi retractor is used during Cesarean sections, when compared to traditional pannus retractor techniques, montogmery straps.
Time Frame: 24 hours from placement of device
Population: Patient data not collected
Arm/Group | Treatment | Standard
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Duration of Surgery or Length of Time From Skin Incision to Delivery of the Infant
Description: To determine if there is a difference in duration of surgery or length of time from skin incision to delivery of the infant between the treatment group and the control/standard group.
Time Frame: At time of surgery
Population: Data were not collected.
Arm/Group | Treatment | Standard
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Hemoglobin
Description: To determine if there is a difference in change in hemoglobin between the control/standard group and the treatment group.
Time Frame: 24 hours after surgery
Population: Data were not collected
Arm/Group | Treatment | Standard
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Estimated Blood Loss
Description: To determine if there is a difference in estimated blood loss between the treatment group and the control/standard group.
Time Frame: At time of surgery
Population: Data were not collected.
Arm/Group | Treatment | Standard
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Postoperative Length of Stay
Description: To determine if there is a difference in postoperative length of stay between the treatment group and the control/standard group.
Time Frame: 3-4 days
Population: Data were not collected.
Arm/Group | Treatment | Standard
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Other Complication Rate
Description: To determine if there is a difference in other complication rates between the treatment group and the control/standard group.
Time Frame: 6 weeks
Population: Data were not collected.
Arm/Group | Treatment | Standard
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Need for Hospital Readmission or Emergency Room Visits
Description: To determine if there is a difference in need for hospital readmission or emergency room visits between the treatment group and the control/standard group.
Time Frame: 6 weeks
Population: Data were not collected.
Arm/Group | Treatment | Standard
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Other (Not Including serious) adverse events were not monitored/assessed
Arm/Group | Treatment | Standard
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No